CLINICAL TRIAL: NCT01626365
Title: The Effect of Double-lumen Tube Thermosoftening Before Intubation to Reduce Hoarseness and Sore Throat
Brief Title: Thermosoftening of Double-lumen Tube to Reduce Sore Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHBahk_DLT_thermosoftening
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Hoarseness; Sore Throat; Vocal Cord Injuries
Keywords: double-lumen tube; intubation; thermosoftening
MeSH Terms: conditions — Hoarseness; Pharyngitis

ARMS (2):
- non-thermosoftening (Active Comparator): Double-lumen tube is put into a bottle of normal saline at room temperature (25°C) before intubation.
  Interventions: Procedure: non-thermosoftening
- thermosoftening (Experimental): Double-lumen tube is put into a bottle of warm normal saline (40°C) before intubation.
  Interventions: Procedure: thermosoftening

INTERVENTIONS:
Procedure: non-thermosoftening — Intubation is performed with a double-lumen tube put into normal saline at room temperature.
  Arms: non-thermosoftening
Procedure: thermosoftening — Intubation is performed with a double lumen tube put into warm normal saline (40°C).
  Arms: thermosoftening

SUMMARY:
The purpose of this study is to investigate the effect of double-lumen tube thermosoftening before intubation to reduce postoperative hoarseness and sore throat.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic surgery that require the placement of left-sided double-lumen tubes

Exclusion Criteria:

* Preoperative hoarseness or sore throat
* History of upper airway diseases
* Anticipated difficult airway
* Anesthesia time longer than 6 hours

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Postoperative hoarseness | up to 3 days after surgery
postoperative sore throat | up to 3 days after surgery

SECONDARY OUTCOMES:
Vocal cord injuries | up to 1 day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Seo JH, Cho CW, Hong DM, Jeon Y, Bahk JH. The effects of thermal softening of double-lumen endobronchial tubes on postoperative sore throat, hoarseness and vocal cord injuries: a prospective double-blind randomized trial. Br J Anaesth. 2016 Feb;116(2):282-8. doi: 10.1093/bja/aev414. PMID 26787799